CLINICAL TRIAL: NCT06610929
Title: Metabolites From the Intestinal Microbiota and Visceral Pain Associated With Chronic Intestinal Pseudo-obstruction (CIPO) in Children
Brief Title: Intestinal Microbiota and Visceral Pain in Chronic Intestinal Pseudo-Obstruction Syndrome (CIPO)
Acronym: METADOLOMIC
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240437; IDRCB: 2024-A00717-40 (Registry Identifier: ANSM)
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Intestinal Obstruction
Keywords: Microbiota
MeSH Terms: conditions — Intestinal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Digestive effluent
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic Intestinal Pseudo-Obstruction Syndrome (CIPO) is a rare gastrointestinal motility disorder. CIPO evolves through iterative flare-ups that can be triggered by viral or bacterial infections, psychological stress, or malnutrition. All of these factors are associated with dysbiosis of the intestinal microbiota (IM). Many studies have associated visceral pain with dysbiosis of the IM, particularly in the context of irritable bowel syndrome (IBS), a painful pathology associated with transit disorders. The team in Dr. Cénac's laboratory has demonstrated the analgesic effect of a bacterial lipid produced by an intestinal bacterium in the context of IBS. The study hypothesize that CIPO patients have a taxonomic and functional dysbiosis of the IM responsible for hyperactivation of sensory neurons inducing visceral pain.

DETAILED DESCRIPTION:
The aim of the study is to identify metabolites differentially produced by the gut microbiota of CIPO patients with visceral pain to determine their effect on the host with a focus on intestinal homeostasis.

For that, 3 samples of digestive effluent will be collected in paediatric CIPO patients.

Then, the study will:

1. Characterize the intestinal microbiota of digestive effluents from painful and non-painful pediatric CIPO patients.
2. Quantify bacterial lipids in digestive effluents from painful and non-painful paediatric CIPO patients. In ileal effluents, we will perform absolute quantification of the bacterial lipidome. We will quantify short-chain fatty acids by gas chromatography coupled with mass spectrometry and, long-chain beta-hydroxylated fatty acids, GABA-lipopeptides, lipoamines and primary and secondary bile acids by liquid chromatography coupled with tandem mass spectrometry.
3. Test the function of these bacterial lipids on sensory neuronal activity in a primary culture of mouse dorsal root ganglia. The effects of bacterial lipids on sensory neurons will be evaluated in a primary culture of mouse dorsal root ganglia. We will quantify calcium mobilization in sensory neurons treated with the lipid compounds identified above. In a second step, in order to determine their inhibitory potential, the same experiments will be performed on neurons activated by a calcium channel receptor agonist, TRPV1 (capsaicin) or by a mix of agonists (histamine, serotonin and bradykinin) of G protein-coupled receptors involved in visceral hypersensitivity

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 1 to 21 years
* Patient diagnosed with CIPO for at least 12 months (= patients meeting at least 2 of the following 4 criteria: 1. Recurrent episodes of intestinal dilatation, 2. Inability to maintain nutrition, 3. Intestinal neuromuscular alteration and 4. Genetic variants.)
* Patient with an ileal or colonic digestive diversion
* Signature of informed consent by both holders of parental authority and agreement in principle given orally by the subject;
* Patients affiliated to a social security scheme

Exclusion Criteria:

-

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient diagnosed with CIPO for at least 12 months (= patients meeting at least 2 of the following 4 criteria: 1. Recurrent episodes of intestinal dilatation, 2. Inability to maintain nutrition, 3. Intestinal neuromuscular alteration and 4. Genetic variants.)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Nature and quantity of bacteria identified by sequencing in the digestive effluent of painful and non-painful CIPO pediatric patients | 12 months
  microbiota analysis by DNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Alexis MOSCA, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France